CLINICAL TRIAL: NCT05326243
Title: A Phase 1/2 Multicenter, Open-label, Single-arm Study to Evaluate the Safety and Efficacy of CD19-targeted Chimeric Antigen Receptor T-cell (CD19 CAR-T; PL001) Therapy in Patients With Relapsed or Refractory B-cell Lymphoma
Brief Title: Phase 1/2 Study of CD19 Chimeric Antigen Receptor T-cell (CD19 CAR-T; PL001) for Relapsed or Refractory B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pell Bio-Med Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL001-NHL-201
Record Dates: First submitted 2022-03-25; First posted 2022-04-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Diffuse Large B Cell Lymphoma; Primary Mediastinal Large B Cell Lymphoma; Large B-cell Lymphoma; Follicular Lymphoma Grade 3A; Follicular Lymphoma Grade 3B
Keywords: DLBCL; PMLBCL; FL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: This study is a multiple-center, non-randomized, open-label, phase 1/2 study. Lymphodepletion chemotherapy (intravenous infusion of fludarabine plus cyclophosphamide will be administered for 3 consecutive days before the day of PL001 dosing (Day 0) and should take place within Day -5 to Day -3 (a safe window for a small subset of patients will be D -7 to D -3). This study will test two dose levels of PL001, dose level 1 and dose level 2. In Phase 1, doses will be tested in the modified "3 + 3" design initiating with dose level 1. The primary objective of Phase 1 is to assess the safety of PL001 and find the recommended phase 2 dose. Phase 2 expansion cohort will receive PL001 at the recommended dose determined in Phase 1. Efficacy evaluations using computed tomography (CT) and positron emission tomography (PET) will be performed at 1, 3, 6, 9, and 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19-targeted chimeric antigen receptor T-cell (Experimental): Patients will receive a lymphodepletion chemotherapy with fludarabine plus cyclophosphamide for three consecutive days(Day -5 to Day -3) before infusion of CD19-targeted chimeric antigen receptor T-cell (CD19 CAR-T). Patients will receive the CD19 CAR-T(also known as PL001) infusion on Day 0.
  Interventions: Biological: CD19-targeted chimeric antigen receptor T-cell

INTERVENTIONS:
Biological: CD19-targeted chimeric antigen receptor T-cell — Drug: Fludarabine
  patients will receive a lymphodepletion chemotherapy with Fludarabine 25 mg/m2/day IV for 3 days on Day-5 to Day-3(a safe window for a small subset of patients will be D -7 to D -3).
  Drug: Cyclophosphamide
  patients will receive a lymphodepletion chemotherapy with cyclophosphamide 300 mg/m2/day IV for 3 dys Day-5 to Day-3(a safe window for a small subset of patients will be D -7 to D -3).
  Biological: CD19 CAR-T
  CD19 CAR-T cells will be administered using as a single dose at 0.1-9*10^6 cells/kg on Day 0 after completion of the lymphodepletion chemotherapy. The body weight calculated for PL001 dose is the actual body weight on the day of leukapheresis.
  Other Names: PL001

SUMMARY:
This is a multiple center, non-randomized, open-label, phase 1/2 study. The primary objective of Phase 1 is to evaluate the safety of PL001 and find the recommended Phase 2 dose (RP2D). The objective of Phase 2 is to evaluate the safety and efficacy of CD19 CAR-T(known as PL001).

DETAILED DESCRIPTION:
Cluster of differentiation (CD) 19 chimeric antigen receptor T-cell (CAR-T) has been a very promising treatment option for multiple types of B-cell lymphoma. Kymriah® (tisagenlecleucel, Novartis) and Yescarta® (axicabtagene ciloleucel, Gilead) were licensed by the United States Food and Drug Administration (US FDA) and European Medicines Agency (EMA) in 2017 to treat relapsed or refractory B-cell acute lymphoblastic leukemia (B-ALL), diffuse large B-cell lymphoma (DLBCL), and High-grade B-cell lymphoma (HGBCL). A third anti-CD19 CAR-T product, Tecartus (brexucabtagene autoleucel, Gilead) was approved by the US FDA for relapsed and refractory mantle cell lymphoma (MCL) in July 2020. In February 2021, another product, Breyanzi® (lisocabtagene maraleucel, Juno Therapeutics, Inc.), was approved by the US FDA for relapsed or refractory large B-cell lymphoma after two or more lines of systemic therapy, including DLBCL not otherwise specified (including DLBCL arising from indolent lymphoma), high-grade B-cell lymphoma, Primary mediastinal large B cell lymphoma (PMLBCL), and Gr. 3b FL.

Currently, in Taiwan, no CD19 CAR-T therapies are available commercially.This Phase 1/Phase 2 study will test PL001, a CD19 CAR-T therapy manufactured by Pell Bio-Med Technology Co., Ltd., as a monotherapy for relapsed or refractory B-cell lymphoma. The Phase 1 of the study will be conducted to establish a dose range that is well tolerated by the majority of patients and to provide a safety profile of PL001 in the target patient population. The results of the Phase 1 of the study will recommend the dose selection for the Phase 2 of the study. Phase 2 of the study will assess the efficacy and safety of PL001 in patients with relapsed or refractory B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Screening 1:

1. Patient is ≥14 years of age, inclusive, at the time of signing the informed consent.
2. Histologically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMLBCL), large B-cell lymphoma transformed from follicular lymphoma (FL), or grade 3a or 3b FL.
3. On-site documentation of CD19 on the dominant population of cancer cells.
4. Disease status should meet any one of the below:

   1. Patients with previous autologous-hematopoietic stem cell transplantation (auto HSCT) have relapsed, progressive, or refractory disease (defined as having not achieved a CR) after transplantation regardless of lines of systemic therapy.
   2. Patients without previous HSCT have relapsed, progressive, or refractory disease (defined as having not achieved a CR) after at least 2 lines of systemic therapy, including anti-CD20 antibody and anthracycline.
5. Have no available effective systemic therapy as judged by the Investigator.
6. At least one measurable non-CNS (central nervous system) lesion based on Lugano classification for lymphoma.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
8. Life expectancy of at least 3 months.
9. Patient is male or female.
10. A male patient must agree to use a highly effective contraception as detailed in Section 10.4 (Appendix 4) during the treatment period and for at least 2 years after the dose of PL001 and refrain from donating sperm during this period.

    Female Patients:
11. A female patient is eligible to participate if she is not pregnant (Section 10.4; Appendix 4), not breastfeeding, and at least one of the following conditions applies:

    • Not a woman of childbearing potential (WOCBP) as defined in Section 10.4 (Appendix 4).

    OR

    • A WOCBP who agrees to follow the contraceptive guidance in Section 10.4 (Appendix 4) during the treatment period and for at least 2 years after the dose of PL001 and refrain from donating ova during this period.
12. Patient/patient's parent/legal guardian is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Screening 2:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
2. CAR-T is successfully manufactured and ready for use, from cells harvested by non mobilized leukapheresis.
3. WOCBP who have a negative serum pregnancy test at Screening 2.

Exclusion Criteria:

Screening 1:

1. Chronic lymphocytic leukemia with Richter's transformation.
2. Primary CNS lymphoma. (Non-primary CNS lymphoma with CNS involvement is eligible).
3. Primary intra-ocular lymphoma.
4. Prior CD19 targeted therapy, such as CAR-T, Bi-specific T-cell engagers (BiTE), or monoclonal antibody.
5. History of cancers (includes myelodysplastic syndrome) other than non-melanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast) unless disease-free without active treatment for at least 3 years.
6. History of allogeneic HSCT.
7. History of autologous HSCT within 3 months prior to consent.
8. Received any investigational product within 4 weeks prior to consent.
9. Systemic anticancer therapy within 3 weeks prior to apheresis.
10. Long-term use of systemic corticosteroids, defined as daily use >10 mg of prednisolone or equivalent, within 2 weeks prior to leukapheresis.

    Exception examples:
    * Nasal, ophthalmic, inhaled, intra-articular, and topical steroid preparation.
    * Short term systemic steroid for drug, contrast, or blood transfusion allergic reaction management.
    * Low dose maintenance steroid therapy for other conditions (e.g., asthma).
11. Use of long-acting and short-acting myeloid growth factor within 2 weeks, 5 days prior to leukapheresis, respectively.
12. Received anti-thymocyte globulin within 4 weeks prior to consent.
13. Intrathecal chemotherapy within 1 week prior to leukapheresis.
14. Inadequate major organ functions at Screening, which were defined as any of below:

    1. absolute neutrophil count (ANC) <500/µL
    2. Absolute lymphocyte count (ALC) <300/µL, excluding leukemic cells.
    3. Hemoglobin (Hb) <8.0 g/dL
    4. Platelet count <75,000/µL without transfusion support within 3 days
    5. e. Baseline O2 saturation <92% by pulse oximetry at room air
    6. Significant CNS diseases such as dementia, major stroke, seizure while under antiepileptic drug
    7. Aspartate aminotransferase (AST) >5 × upper limit of normal (ULN) and alanine aminotransferase (ALT) >5 × ULN, or total bilirubin >2 × ULN (except for constitutional jaundice)
    8. Serum creatinine > 1.5 × ULN and estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m², as calculated by the Cockcroft-Gault formula.
    9. Significant cardiac disease including but not limited to: left ventricular ejection fraction (LVEF) <50%, QTc(the corrected QT interval) > 480 msec based on Fredericia's formula, clinically significant arrhythmias, history of myocardial infarction or unstable angina within 3 months prior to consent.
15. Active hepatitis B virus (HBV) infection defined as detectable HBV DNA (Patients with positive anti-hepatitis B core antibody [HBcAb] must consent to regular monitoring of HBV DNA, and anti-HBV prophylaxis with oral anti-viral agent (such as entecavir) is mandatory until End-of-Study visit [Visit 15].)
16. Active hepatitis C virus (HCV) infection defined as positive anti- HCV antibody plus detectable HCV RNA.
17. Positive for human immunodeficiency virus (HIV) or human T-cell lymphotropic virus (HTLV) infection.
18. Uncontrolled acute life-threatening bacterial, viral, or fungal infection (e.g., the need for intravenous therapeutic antibiotics, blood culture positive ≤72 hours prior to apheresis).

21. Any medical conditions which might compromise the patient's safety from leukapheresis, lymphodepletion chemotherapy, or CAR-T therapy and anticipated AEs, according to the Investigator's evaluation.

22.Patients with insufficient leukapheresis cells.

Screening 2:

1. Inadequate major organ functions at Screening which were defined as any of below:

   1. ANC <500/µL
   2. Hb <8.0 g/dL
   3. Platelet count <50,000/µL, without transfusion support within 3 days
   4. Baseline O2 saturation <92% by pulse oximetry on room air
   5. AST >5 × ULN and ALT>5 × ULN, or total bilirubin >2 × ULN (except for constitutional jaundice)
   6. Significant CNS diseases such as dementia, major stroke, seizure while under antiepileptic drug
   7. Serum creatinine > 1.5 × ULN and estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m², as calculated by the Cockcroft-Gault formula.
2. Long-term use of systemic corticosteroids, defined as daily use >10 mg of prednisolone or equivalent.

   Exception examples:
   * Nasal, ophthalmic, inhaled, intra-articular, and topical steroid preparation.
   * Short term systemic steroid for drug, contrast, or blood transfusion allergic reaction management.
   * Low dose maintenance steroid therapy for other conditions (e.g., asthma).
3. Use of long-acting and short-acting myeloid growth factor within 12 days, 2 days prior to lymphodepletion therapy, respectively.
4. Uncontrolled acute life-threatening bacterial, viral, or fungal infection (e.g. the need for intravenous therapeutic antibiotics, blood culture positive ≤72 hours prior to lymphodepletion).
5. Any medical condition which might compromise the patient's safety because of lymphodepletion chemotherapy or CAR-T therapy and anticipated AEs, according to the Investigator's opinion.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose-limiting toxicities | 30 days
  Dose-limiting toxicities through 30 days after PL001 infusion
Phase 2: best overall response (BOR) | 12 months
  The best overall response (BOR) comprising patients with partial and complete responses according to Lugano criteria assessed based on the image review result provided by the Independent Central Review from the start of infusion of PL001 until next subsequent cancer-specific therapy, disease progression, death, or end of study, whichever comes first

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Treatment-related adverse events | 12 months
  Treatment-related adverse events assessed by CTCAE v 5.0. Overall grading of Cytokine Release Syndrome, immune effector cell associated neurotoxicity syndrome, based on the American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Phase 1 and Phase 2: Best overall response (BOR) | 12 months
  The BOR of patients with partial and complete responses according to Lugano criteria assessed by the Investigator.
Phase 1 and Phase 2: Median duration of response (mDOR) | 12 months
  Median duration of response (mDOR) measured from the time of initial documented response (complete response or partial response) until documented disease progression or death.
Phase 1 and Phase 2: Progression-free survival (PFS) | 12 months
  Progression-free survival (PFS) defined as the time from the infusion of PL001 until objective disease progression or death, whichever occurs first.
Phase 1 and Phase 2: Overall survival (OS) | 12 months
  Overall survival (OS) defined as the time from the infusion of PL001 until death from any cause.
Phase 1 and Phase 2: the health-related quality of life (HRQoL) | 12 months
  Change in the health-related quality of life (HRQoL) by FACT-Lym (the Functional Assessment of Cancer Therapy-Lymphoma)® version 4

OTHER OUTCOMES:
Phase 1 and Phase 2: Pharmacokinetic (PK) profile of PL001-Persistence of PL001 by flow cytometry | 12 months
  Persistence of PL001 in peripheral blood using flow cytometry
Phase 1 and Phase 2: Pharmacokinetic (PK) profile of PL001-Persistence of PL001 by qPCR | 12 months
  PL001 transgene levels by qPCR (quantitative polymerase chain reaction) in peripheral blood
Phase 1 and Phase 2: Quality assurance of the product | [From start of CAR-T manufacturing to CAR-T infusion, estimated to be 45 days]
  Rates for successful production and infused patients
Phase 1 and Phase 2: To assess the cytokine biomarkers | 12 months
  Cytokine concentrations in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Lung Lin, MD, Study Chair — Pell Bio-Med Technology Co., Ltd.
Locations (5):
- Taiwan (5):
  - National Taiwan University Hospital, Taipei, Taiwan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chi Mei Medical Center, Tainan
  - Taipei Medical University - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No